CLINICAL TRIAL: NCT05015088
Title: Effectiveness of Gastrocnemius Stretching
Acronym: Gastroc
Status: Completed | Type: Observational
Sponsor: Regis University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Stephanie Albin, Principal Investigator, Regis University
Other Study IDs: COMIRB
Record Dates: First submitted 2021-08-11; First posted 2021-08-20 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Gastrocnemius Tightness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastrocnemius Stretching Group: The study will enroll 20 healthy subjects between the ages of 18 to 65 years old. Individuals will be recruited from multiple locations. Exclusion criteria include: any boney or tendinous foot/ankle operative procedure, diagnosis of neuromuscular disorder, any previous ankle fracture or degenerative changes that would limit dorsiflexion range of motion. Participants must have no obvious gait asymmetries demonstrated through observation. In addition, participants who are pregnant will be excluded from participation in the study.
  Interventions: Other: No interventions will be performed in this study

INTERVENTIONS:
Other: No interventions will be performed in this study — This study will not include any intervention

SUMMARY:
The aims of this study are to: (1) determine muscle activation of the tibialis posterior muscle during different common gastrocnemius stretches and (2) radiographically quantify the tibial-calcaneal angle during the common stretching positions. We hypothesize that stretching over the edge of a step with the arch supported will minimize the activation of the tibialis posterior muscle in addition to increasing the tibial-calcaneal angle.

DETAILED DESCRIPTION:
Many studies have assessed the effect of dynamic and passive support of the medial longitudinal arch. The posterior tibial tendon is the main dynamic stabilizer of the medial longitudinal arch, although peroneus/fibularis longus, flexor digitorum longus, and flexor hallucis longus also contribute to a lesser degree. Passive structures also a play role in supporting the arch and include the plantar fascia, plantar ligaments and spring ligament. These plantar structures aid in preventing collapse of the arch during weight bearing.

Several studies have demonstrated that increased tension from the triceps surae can lead to flattening of the arch. Gastrocnemius muscle tightness in particular is thought to be partially responsible for many forefoot and midfoot conditions in non-neurologically impaired patients. Therefore, identifying effective ways to stretch the gastrocnemius muscle without creating increased stress through dynamic structures that support the longitudinal arch may be important for the management of individuals with limited gastrocnemius flexibility.

Common ways to stretch the gastrocnemius include a runner's stretch, stretching with the foot fully supported on a ramp, stretching with the arch of the foot supported on the edge of step and the heel dropping down toward the ground and lastly, stretching with the ball of the foot supported on the edge of a step and the heel dropping down toward the ground. To our knowledge no other studies have assessed the muscle activation of the tibialis posterior muscle via indwelling EMG activation in addition to radiographic measurements to determine the effectiveness of common gastrocnemius stretches. Therefore, the aims of this study are to determine muscle activation of the tibialis posterior muscle during different common gastrocnemius stretches and to radiographically quantify the tibial-calcaneal angle. We hypothesize that stretching over the edge of a step with the arch supported will minimize the activation of the tibialis posterior muscle in addition to increasing the tibial-calcaneal angle more than the other stretching positions.

ELIGIBILITY:
Inclusion Criteria:

• 20 healthy subjects between the ages of 18 to 65 years old.

Exclusion Criteria:

* any boney or tendinous foot/ankle operative procedure
* diagnosis of neuromuscular disorder
* any previous ankle fracture or degenerative changes that would limit dorsiflexion range of motion
* no obvious gait asymmetries demonstrated through observation
* participants who are pregnant will be excluded from participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
EMG activation | up to 6 months
  EMG activation of tibialis posterior muscle during 4 common gastrocnemius stretching positions
Radiographic evaluation | up to 6 months
  radiographically the angle of the tibia-calcaneus axis and calcaneal pitch between four different common gastrocnemius stretches

SECONDARY OUTCOMES:
Relationship between foot posture and radiographic evaluation of tibia-calcaneal angle | up to 6 months
  Assess if there is a relationship between radiographic stretching position and foot posture

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Albin, PhD, Principal Investigator — Regis University
Locations (1):
- Regis University, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mueller TJ. Acquired flatfoot secondary to tibialis posterior dysfunction: biomechanical aspects. J Foot Surg. 1991 Jan-Feb;30(1):2-11. PMID 2002182
- [Background] Thordarson DB, Schmotzer H, Chon J, Peters J. Dynamic support of the human longitudinal arch. A biomechanical evaluation. Clin Orthop Relat Res. 1995 Jul;(316):165-72. PMID 7634700
- [Background] Huang CK, Kitaoka HB, An KN, Chao EY. Biomechanical evaluation of longitudinal arch stability. Foot Ankle. 1993 Jul-Aug;14(6):353-7. doi: 10.1177/107110079301400609. PMID 8406252
- [Background] DiGiovanni CW, Kuo R, Tejwani N, Price R, Hansen ST Jr, Cziernecki J, Sangeorzan BJ. Isolated gastrocnemius tightness. J Bone Joint Surg Am. 2002 Jun;84(6):962-70. doi: 10.2106/00004623-200206000-00010. PMID 12063330
- [Background] Maeda N, Komiya M, Nishikawa Y, Morikawa M, Tsutsumi S, Tashiro T, Fukui K, Kimura H, Urabe Y. Effect of Acute Static Stretching on the Activation Patterns Using High-Density Surface Electromyography of the Gastrocnemius Muscle during Ramp-Up Task. Sensors (Basel). 2021 Jul 15;21(14):4841. doi: 10.3390/s21144841. PMID 34300581